Comparison of Flexor Hallicus Brevis and Adductor Pollicis as Sites for Neuromuscular Monitoring With Electromyography (Thumb vs Great Toe) After Sugammadex Administration

NCT04312256

1/15/2021

# Comparison of Flexor Hallucis Brevis and Adductor Pollicis Muscles (Thumb vs. Great Toe) as Sites for Neuromuscular Monitoring with Electromyography after Sugammadex Antagonism

Regulatory Sponsor Principal Investigator: J. Ross Renew, MD

Funding Sponsor: Departmental Resources

**Protocol Number:** IRB # 19-011705

Study Product: TetraGraph

**Initial version:**[10Jan2020] Version (1.0)

Revision: [02Dec2020] Version (2.0)

[14Dec2020] Version (2.1) [15Jan2021] Version (3.0)

# **Table of Contents**

| 1 | P | PROTOCOL APPROVAL FORM | 4 |
|---|---|---|---|
| 2 | L | JST OF ABBREVIATIONS | 5 |
| 3 | S' | TUDY SUMMARY | 6 |
| 4 | | NTRODUCTION | |
| • | 4.1<br>4.2<br>4.3 | ABSTRACT | 7<br>7 |
| 5 | _ | TUDY OBJECTIVES | |
| | | TUDY DESIGN | |
| 6 | 6.1<br>6.2<br>6.3<br>6.4<br>6.5<br>6.6 | GENERAL DESCRIPTION NUMBER OF SUBJECTS DURATION OF PARTICIPATION PRIMARY STUDY ENDPOINTS SECONDARY STUDY ENDPOINTS IDENTIFICATION OF SOURCE DATA | 10<br>10<br>10<br>11 |
| 7 | S | SUBJECT SELECTION ENROLLMENT AND WITHDRAWAL | 12 |
| | | INCLUSION CRITERIA EXCLUSION CRITERIA SUBJECT RECRUITMENT, ENROLLMENT AND SCREENING EARLY WITHDRAWAL OF SUBJECTS 4.1 When and How to Withdraw Subjects 4.2 Data Collection and Follow-up for Withdrawn Subjects | 12<br>12<br>12 |
| 8 | S' | TUDY DEVICE | 13 |
| | 8.1<br>8.2<br>8.3 | DESCRIPTION | 13 |
| 9 | S' | TUDY PROCEDURES | 14 |
| | 9.1<br>9.2<br>9.3 | VISIT 1 (SCREENING AND ENROLLMENT UP TO THE DAY OF SURGERY) VISIT 2 (RANDOMIZATION AND TREATMENT – DAY OF SURGERY) SCHEDULE OF EVENTS | 14 |
| 10 | S' | TATISTICAL PLAN | 15 |
| | 10.1<br>10.2<br>10.3 | STATISTICAL METHODS | 15 |
| 11 | <b>S</b> . | SAFETY AND ADVERSE EVENTS | 16 |
| | 1. | DEFINITIONS | 16<br>16 |

| 11. | .1.4 Adverse Event Reporting Period | 17 |
|-------|----------------------------------------------------------------|----|
| 11. | .1.5 Preexisting Condition | |
| 11. | .1.6 Post-study Adverse Event | |
| 11. | .1.7 Hospitalization, Prolonged Hospitalization or Surgery | 17 |
| 11.2 | RECORDING OF ADVERSE EVENTS | |
| 11.3 | REPORTING OF SERIOUS ADVERSE EVENTS AND UNANTICIPATED PROBLEMS | 18 |
| 11. | .3.1 Sponsor-Investigator reporting: notifying the Mayo IRB | 18 |
| 11.4 | MEDICAL MONITORING | 20 |
| 12 DA | ATA HANDLING AND RECORD KEEPING | 20 |
| 12.1 | Confidentiality | 20 |
| 12.2 | Source Documents | 20 |
| 12.3 | CASE REPORT FORMS | |
| 12.4 | Data Management | |
| 12.5 | Data Processing | |
| 12.6 | DATA SECURITY AND CONFIDENTIALITY | |
| 12.7 | DATA QUALITY ASSURANCE | 21 |
| 12.8 | DATA CLARIFICATION PROCESS | |
| 12.9 | RECORDS RETENTION | |
| 13 ST | TUDY MONITORING, AUDITING, AND INSPECTING | 22 |
| 13.1 | STUDY MONITORING PLAN | 22 |
| 13.2 | AUDITING AND INSPECTING | 22 |
| 14 ET | THICAL CONSIDERATIONS | 22 |
| 15 ST | TUDY FINANCES | 22 |
| 15.1 | Funding Source | 22 |
| 15.1 | Conflict of Interest. | |
| 15.3 | SUBJECT STIPENDS OR PAYMENTS | |
| | JBLICATION PLAN | |
| 17 RI | EFERENCES | 23 |
| 18 LI | ST OF IN-TEXT TABLES | 25 |
| 18.1 | SCHEDULE OF EVENTS | 25 |
| 18.2 | Intraoperative Data | 25 |
| 18.3 | MONITORING DATA | 26 |
| 19 LI | ST OF IN-TEXT FIGURES | 28 |
| 19.1 | TetraGraph | 28 |
| 17.1 | * £ 1.4. • 1.4. 1.1. 1.1. 1.1. 1.1. 1.1. 1. | |

# 1 Protocol Approval Form

Protocol Number: 19-011705

Study Name: Comparison of Flexor Hallucis Brevis and Adductor Pollicis Muscles (Thumb vs Great Toe) as Sites for Neuromuscular Monitoring with Electromyography after Sugammadex Antagonism

This protocol has been reviewed and approved by the following:

I Line

J. Ross Renew, MD Principal Investigator 01/15/2021

#### 2 List of Abbreviations

AE Adverse Event/Adverse Experience

AMG Acceleromyography
CE Conformite Europeene
CFR Code of Federal Regulations

cMAPs Compound Muscle Action Potentials

CRF Case Report Form

CTSA Center for Translational Science Activities

DSMB Data and Safety Monitoring Board

EHR Electronic Health Record

EMG Electromyography

FDA Food and Drug Administration

GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

IB Investigator's Brochure ICU Intensive Care Unit

IRB Institutional Review Board

KMG Kinemyography MMG Mechanomyography

NMBA Neuromuscular Blocking Agent

Non-UPIRTSO Non-Unanticipated Problems Involving Risk to Subjects or

Others

PACU Post Anesthesia Care Unit PHI Protected Health Information

PI Principal Investigator

SAE Serious Adverse Event/Serious Adverse Experience

SGX Sugammadex

SOP Standard Operating Procedure

TOF Train-of-four TOFC Train-of-four count TOFR Train-of-four ratio

UPIRTSO Unanticipated Problems Involving Risk to Subjects or Others

VNRS Verbal Numeric Rating Scale

# 3 Study Summary

| Title | Comparison of Flexor Hallucis Brevis and Adductor Pollicis Muscles (Thumb vs Great Toe) as Sites for Neuromuscular Monitoring with Electromyography after Sugammadex Antagonism |
|---|---|
| Running Title | Thumb vs Great Toe Recovery |
| Phase | N/A |
| Methodology | Randomized, Open-Label |
| Overall Study<br>Duration | 12 months |
| Subject Participation<br>Duration | 2 to 5 hours |
| Single or Multi-Site | Single site |
| Objectives | The primary aim of this study is to assess the onset of neuromuscular blockade and recovery profiles of aminosteroidal NMBAs after sugammadex at the flexor hallucis brevis and adductor pollicis muscles |
| Number of Subjects | 130 |
| Diagnosis and Main<br>Inclusion Criteria | Patients undergoing elective surgery and requiring administration of aminosteroidal NMBAs (rocuronium, vecuronium) intraoperatively |
| Study Device | TetraGraph |
| Duration of<br>Administration | Single stimulation of flexor hallucis brevis and adductor pollicis muscles repeated at specific intervals as outlined in the Study Procedures (Section 9.2) |

#### 4 Introduction

This document is a protocol for a human research study. This study will be carried out in accordance with the applicable United States government regulations and Mayo Clinic research policies and procedures.

#### 4.1 Abstract

Residual neuromuscular blockade is a common occurrence in the post-anesthesia care unit (PACU) when neuromuscular blocking agents (NMBAs) have been used in the operating room. The only method of reliably detecting residual neuromuscular blockade is through the use of quantitative neuromuscular monitors. Unfortunately, several barriers exist that have prevented the widespread use of these devices. For instance, there is a paucity of quantitative neuromuscular monitors commercially available. Also, two modalities of quantitative monitoring, kinemyography and acceleromyography, rely on movement of the muscles of interest, a characteristic frequently compromised during patient positioning for surgical procedures in which the patient's arms are secured under surgical drapes (laparoscopic, bariatric, robotic, spine, and neurosurgical procedures) or in uncooperative awake patients in the PACU or intensive care unit (ICU). The aim of this investigation is to determine the different muscle sensitivities to NMBA and reversal agents by comparing responses at two different monitoring sites as measured with a new quantitative monitor. The TetraGraph (Senzime AB, Uppsala, Sweden) is a standalone electromyography (EMG)-based quantitative monitor that recently received Conformité Européene (CE) and US Food and Drug Administration (FDA) approvals. EMG measures electrical activity within the muscle following peripheral nerve stimulation, and is unaffected by involuntary patient motion or by restricted muscle movements from surgical positioning. We plan to compare measurements obtained with two Tetragraph devices, one monitoring the adductor pollicis (thumb) muscle and the other monitoring the flexor hallucis brevis (great toe) muscle, during onset, maintenance, and recovery of neuromuscular blockade. This will include monitoring every 20 sec for onset of blockade (defined as Train-of-four count, TOFC =0) following rocuronium administration, during maintenance of neuromuscular block as required by surgical conditions, and following reversal administration until adequate recovery is documented (train-of-four ratio, TOFR > 0.9).

# 4.2 Background

Postoperative residual weakness from neuromuscular blockade continues to be a common problem in the post-anesthesia care unit (PACU). Despite the routine use of reversal agents, a significant number of patients continue to arrive in the PACU with objective evidence of residual neuromuscular blockade (Naguib, Kopman, and Ensor 2007; Cammu et al. 2006; Fortier et al. 2015; Renew and Brull 2019). While not every patient with residual weakness develops a postoperative complication, many can develop avoidable critical respiratory events (Murphy et al. 2008; Berg et al. 1997). Furthermore, special populations such as the elderly, are at particular

risk for developing complications related to postoperative residual weakness (Murphy et al. 2015). The use of quantitative monitoring has been demonstrated to reliably reduce the incidence of postoperative residual weakness and the ensuing complications (Todd, Hindman, and King 2014; Todd and Hindman 2015; Murphy et al. 2011). With an abundance of literature supporting the use of objective neuromuscular monitors, a panel of experts recently recommended the universal adoption of such devices whenever NMBA are utilized (Naguib et al. 2018).

Quantitative neuromuscular monitoring devices objectively measure muscle responses and display the results numerically. This is traditionally accomplished by performing a train-of-four (TOF) stimulation at the ulnar nerve and measuring the response of the adductor pollicis muscle. The degree of muscle weakness is determined by calculating the TOF ratio, which consists of the ratio of the fourth muscle contraction to the first (T4/T1). Adequate recovery that excludes clinically significant weakness from neuromuscular blockade is defined as a TOF ratio  $\geq 0.9$ , a measurement that can be determined reliably only with a quantitative monitor (Sundman et al. 2000; Eriksson et al. 1997). Although evidence strongly suggests objective monitors should be used perioperatively whenever NMBAs are administered, these devices can be expensive and require additional training. Many clinicians default to using the antiquated qualitative (subjective) neuromuscular stimulating units such as a peripheral nerve stimulator (PNS) (Grayling and Sweeney 2007; Naguib et al. 2010). The major limitation of PNSs is that they cannot measure the muscle responses (TOFR), and therefore cannot assure complete recovery of muscle strength prior to tracheal extubation and spontaneous respiration.

There are several types of quantitative neuromuscular monitors. These devices can be incorporated into the anesthesia workstation, allowing data to be seamlessly integrated into the electronic medical record. Unfortunately, this setup can preclude using these monitors in the busy OR environment or PACU, as portability is sacrificed. In contrast, other monitors exist as standalone, portable (hand-held) units.

Aside from portability, objective monitors can further be categorized based on the modality utilized to measure responses. Mechanomyography (MMG) measures the force of contraction of the adductor pollicis (thumb) muscle following ulnar nerve stimulation and has served as the traditional "gold-standard." MMG responses are precise and reproducible, however the setup is cumbersome and the lack of commercially available devices has relegated MMG to strictly research purposes. Acceleromyography (AMG) measures acceleration of a muscle group (typically the thumb) in response to stimulation (typically the ulnar nerve). This technique is similar to MMG, but instead of measuring the force of muscle contraction, an accelerometer fixed to the thumb measures the acceleration of the thumb in response to ulnar nerve stimulation. Based on Newton's Second law that states force is proportional to acceleration, the measured acceleration is correlated with the force of contraction in the clinical setting. There are currently two standalone AMG-based monitors available for clinical use: the STIMPOD (Xavant Technologies, Pretoria, South Africa) and the ToFscan (Draeger Medical Inc., Telford, PA).

These devices represent improvements in AMG technology over its predecessor, the TOF-Watch (Schering-Plough Corp., Kenilworth, NJ, USA), as they utilize three-dimensional transducers that can better quantify the complex motion of the thumb. Despite these advances, the use of AMG can be limited due to patient positioning that precludes free motion of the thumb, as well instances of awakening (and uncooperative) patients who may involuntarily move their thumb during measurements, making interpretation of responses impossible. Kinemyography (KMG) is based on similar principles to AMG, and also relies on the thumb being able to move freely. Upon neurostimulation, KMG utilizes a piezoelectric motion sensor that is bent between the thumb and index fingers following muscle contraction. The degree of this bending is quantified and used to determine a TOF ratio. While Datex-Ohmeda (Helsinki, Finland) manufactures a KMG device that can be incorporated into the anesthesia work station, there are no currently available standalone KMG devices. Electromyography (EMG) devices measure electrical activity, termed compound muscle action potentials (cMAPs) following nerve stimulation (typically at the adductor pollicis muscle after ulnar nerve stimulation). As EMG measures cMAPs and does not require freely moving thumbs for accurate measurements, many experts have referred to this monitoring modality as the "new gold standard." (Naguib et al. 2018) TetraGraph (Senzime AB, Uppsala, Sweden) is a standalone EMG-based device that recently received Conformité Européene (CE) and US Food and Drug Administration (FDA) approvals. We have previously investigated this device and presented our findings at several annual meetings such as International Anesthesia Research Society (May 2018, May 2017, May 2013), the Society for Technology in Anesthesia (January 2018), and the American Society of Anesthesiologists (October 2017, October 2012), European Society of Anaesthesiology (June 2018, June 2015). Furthermore, we have submitted abstracts to the PostGraduate Assembly in Anesthesiology in December 2018 as well as a manuscript describing a multi-center, volunteer study investigating TetraGraph versus AMG-based monitors. Our work thus far has found this device to be easy to apply, reliable, and able to provide comparable measurements to other quantitative monitors.

Utilizing recommendations from the Good Clinical Research Practice (GCRP) Guidelines for monitoring of neuromuscular function (Fuchs-Buder et al. 2007), we will investigate the performance of the TetraGraph at two muscle groups: adductor pollicis and flexor hallucis brevis. Specifically, the time points of interest will include the onset of blockade (Train-of-four count =0), maintenance of neuromuscular block as clinically indicated by surgical needs, and recovery from rocuronium blockade with sugammadex, and every 20 seconds following reversal administration until tracheal extubation (as determined by the SOC practice).

#### 4.3 Risks and Benefits

• The benefits of using neuromuscular blockade monitoring devices: Early detection of optimal time for tracheal intubation; optimal management of intraoperative depth of neuromuscular block to facilitate surgical procedures;

determination of appropriate time and dose of sugammadex reversal; and detection of residual neuromuscular blockade

• The risks of using neuromuscular blockade monitoring devices: Slight discomfort when electrical stimulation is administered in awake volunteers; however, our patients will be anesthetized, rendering this risk as extremely minor.

# 5 Study Objectives

# Primary Objective

To compare the time to onset of blockade, level of blockade prior to reversal, and the rate of recovery between flexor hallucis brevis and adductor pollicis muscles following sugammadex administration.

## Secondary Objective

Determine the incidence of postoperative residual weakness at the time of extubation at a center that predominately utilizes quantitative monitoring (defined as TOFR <0.90) and sugammadex.

# 6 Study Design

# 6.1 General Description

This pilot unblinded, single center, prospective, randomized, observational study will involve 130 patients undergoing surgical procedure that requires administration of neuromuscular blocking agents intraoperatively.

# 6.2 Number of Subjects

One hundred twenty

#### 6.3 Duration of Participation

2-5 hours, depending on duration of surgery



# 6.4 Primary Study Endpoints

The primary endpoint of the study will be time of onset of blockade and the rate of recovery following sugammadex administration as recorded simultaneously from the hand (adductor pollicis) and foot (flexor hallucis brevis) muscles.

# 6.5 Secondary Study Endpoints

The secondary endpoint is the incidence of postoperative residual weakness at the time of extubation at a center that predominately utilizes quantitative monitoring (defined as TOFR <0.90) and sugammadex.

#### 6.6 Identification of Source Data

The study data points will be recorded on the developed Case Report Forms (CRFs) by the study team members. In addition to the data collected intraoperatively (<u>Table 18.3</u>), several intraoperative characteristics will also be extracted from the medical record (<u>Table 18.2</u>). These will include type and total dose of NMBA used, time and dose of last NMBA administration, time and dose of specific reversal agent administration, time of tracheal extubation, and TOF ratio at the time of extubation (if available).

# 7 Subject Selection Enrollment and Withdrawal

#### 7.1 Inclusion Criteria

- Age > or = 18 years old
- Patients willing to participate and provide an informed consent
- Patients undergoing an elective surgical procedure that requires use of non-depolarizing NMBA agents administered intraoperatively.
- Patients with planned administration of sugammadex as a neuromuscular blocking reversal agent.

#### 7.2 Exclusion Criteria

- Patients with disorders, such as stroke, carpal tunnel syndrome, broken wrist with nerve damage, Dupuytren contracture, or any similar wrist injury.
- Patients with systemic neuromuscular diseases such as myasthenia gravis
- Patients with significant organ dysfunction that can significantly affect pharmacokinetics of neuromuscular blocking and reversal agents, i.e., severe renal impairment or end-stage liver disease.
- Patients having surgery that would involve prepping the arm or leg into the sterile field

# 7.3 Subject Recruitment, Enrollment and Screening

On a daily basis, there are over 20 elective surgical cases performed at Mayo Clinic in Florida and thus no difficulties in accrual are anticipated based on historical volumes. We will target at least 10 participants per week to complete this study. The initial accrual period will last at least 3 months followed by interim analysis and additional time for accrual will be determined to meet the target. Patients will be provided with a Research Participant Consent and Privacy Authorization Form describing the study devices, protocol, inclusion and exclusion criteria, as well as risks and benefits of participation.

#### 7.4 Early Withdrawal of Subjects

# 7.4.1 When and How to Withdraw Subjects

Patients are free to withdraw at any time and for whatever reason. If patient withdraws consent prior to arrival to operating room, the study data will not be collected. If patient withdraws consent after study data was already completed, the participant will need to provide instructions to the study team to remove his/her data from the data set. Pre-specified reasons for discontinuing include, but are not limited to, the following:

• Patient Request: Patient decided that he/she did not want to continue (for any reason)

• Adverse Event: Patient experienced a related or unrelated event that would interfere with the study objectives/evaluation

- Inclusion/Exclusion Discrepancy/Violation: Patient should not have been enrolled
- Other: Any other reason

#### 7.4.2 Data Collection and Follow-up for Withdrawn Subjects

If a Participant withdraws from the study, no additional attempts will be made to contact the Participant.

# 8 Study Device

## 8.1 Description

TetraGraph device is a FDA approved neuromuscular transmission monitor capable of measuring the depth of neuromuscular block in anesthetized patients who received neuromuscular blocking agents. TetraGraph uses EMG to measure the muscle action potentials that are generated in response to electrical neurostimulation via skin (ECG) electrodes. TetraGraph data is recorded on the monitor's built-in SD card, and all intraoperative data will be recorded and later downloaded for purposes of analysis. The recorded data do not contain PHI, only the date/time of recording, and any additional intraoperative interventions, such as the time of NMBA dose administration, time of antidote administration, time of extubation, etc. These events are flagged in the monitor's integrated SD card recordings.

## 8.2 Method for Assigning Subjects to Treatment Groups

This is an open-label pilot investigation and all study participants are assigned to both standard of care and investigational device use in the operating room. The randomization involves the use of dominant vs non-dominant arm. The placement of the lead on the great toe will correspond with the randomization assignment (if patient's dominant hand is right, and then the right great toe will be used).

The randomization will be performed utilizing REDCap and assigned anesthesia clinical care team will be informed of patients' assigned to guide them with the selection of the assigned treatment option.

#### 8.3 Masking/Blinding of Study

This is an open-label investigation. Masking and blinding procedures are not applicable.

# 9 Study Procedures

## 9.1 Visit 1 (Screening and Enrollment up to the day of surgery)

- Review of medical record
- Informed Consent Patients will be identified during their preoperative appointment and introduced to a study; they will be provided with a copy of the consent document and information about the study. The consenting will take place after additional discussion on the day of surgery.

# 9.2 Visit 2 (Randomization and Treatment – day of surgery)

- Elective surgical procedure as per standard of care
- Anesthetic management will include rocuronium, sevoflurane, and sugammadex at the discretion of the attending anesthesiologist as per standard of care practice.
- Prior to induction of anesthesia, Tetragraph electrodes will be placed over the ulnar nerve and the thumb to measure the response of adductor pollicis, and over the posterior tibial nerve and the great toe to measure the response of the flexor hallucis brevis.
- Following induction of anesthesia but prior to NMBA administration, baseline values will be recorded at both muscle groups after instrument calibration.
- Near the conclusion of the operation but prior to reversal of NMBA, another set of measurements will be taken at both muscle groups.
- Intraoperatively, measurements will be taken every minute until the sugammadex administration, as per usual clinical routine.
- After sugammadex administration, measurements will be taken every 20 seconds until the patient's trachea is extubated.
- Anesthesia providers will be guided on the intraoperative management of neuromuscular block based on the responses recorded from the adductor pollicis muscle, as per usual clinical routine.
- Each neurostimulation with the TetraGraph will be conducted simultaneously by a single study team member.
- Following measurements obtained with both devices at these specified time intervals and assuming TOF ratio is >0.9, the devices will be disconnected and the patient will proceed along the standard recovery pathway.

#### 9.3 Schedule of Events

| | Schedule of Events | |
|-----------------------------|--------------------|---------|
| Study Activity | Visit 1 | Visit 2 |
| Tetragraph | | X |
| Informed consent | X | |
| Review of Medical<br>Record | X | |
| Adverse event evaluation | | X |

#### 10 Statistical Plan

#### 10.1 Sample Size Determination

Based on paired t test, 97 patients will provide 90% power to detect a difference of 0.5 min or larger between hands and feet at 0.05 significance level. A common standard deviation of 1.5 min for hands and feet is assumed based on previous work comparing flexor hallucis brevis and adductor pollicis muscles. However, we will enroll 130 patients to take into account patient loss or missing data. We want to determine a shorter time difference between hand and foot in order to make it applicable in all clinical settings, including rapid sequence induction and intubation.

#### 10.2 Statistical Methods

#### **Descriptive Statistics**

Analysis of agreement between the muscle groups will be compared between the two monitoring sites using the Wilcoxon signed rank test. The limits of agreement are defined as bias  $\pm$  2 SD, where SD denotes the standard deviations of the differences. Limits of agreement are interpreted as the reference range within which 95% of the differences will lie. The bias and the limits of agreements surrounding the bias ( $\pm$  2 SD) will be calculated with 95% confidence intervals. Statistical significance will be defined as a p-value <0.05.

#### **Handling of Missing Data**

This is a prospective pilot study and therefore we do not anticipate any missing data. In the event of any unexpected missing data, no attempt to impute this missing data will be made;

missing data will simply be treated as missing in the statistical analysis, and replacement participants will be enrolled to achieve the target accrual of n=100 participants.

# 10.3 Subject Population(s) for Analysis

Each participant who goes through the surgery and completes monitoring of residual neuromuscular blockade will be included in the primary analysis regardless of study withdrawal for any reason. In the event of any study withdrawals, in secondary analysis we will examine the sensitivity of our results to the exclusion of patients who withdrew.

# 11 Safety and Adverse Events

#### 11.1 Definitions

#### 11.1.1 Unanticipated Problems Involving Risk to Subjects or Others (UPIRTSO)

Any unanticipated problem or adverse event that meets the following three criteria:

- <u>Serious</u>: Serious problems or events that results in significant harm, (which may be physical, psychological, financial, social, economic, or legal) or increased risk for the subject or others (including individuals who are not research subjects). These include: (1) death; (2) life threatening adverse experience; (3) hospitalization inpatient, new, or prolonged; (4) disability/incapacity persistent or significant; (5) birth defect/anomaly; (6) breach of confidentiality and (7) other problems, events, or new information (i.e. publications, DSMB reports, interim findings, product labeling change) that in the opinion of the local investigator may adversely affect the rights, safety, or welfare of the subjects or others, or substantially compromise the research data, **AND**
- <u>Unanticipated</u>: (i.e. unexpected) problems or events are those that are not already described as potential risks in the protocol, consent document, or not part of an underlying disease. A problem or event is "unanticipated" when it was unforeseeable at the time of its occurrence. A problem or event is "unanticipated" when it occurs at an increased frequency or at an increased severity than expected, **AND**
- Related: A problem or event is "related" if it is possibly related to the research procedures.

#### 11.1.2 Adverse Event

An untoward or undesirable experience associated with the use of a medical product (i.e. drug, device, biologic) in a patient or research subject.

#### 11.1.3 Serious Adverse Event

Adverse events are classified as serious or non-serious. Serious problems/events can be well defined and include;

- death
- life threatening adverse experience
- hospitalization

• inpatient, new, or prolonged; disability/incapacity

- persistent or significant disability or incapacity
- birth defect/anomaly

and/or per protocol may be problems/events that in the opinion of the sponsor-investigator may have adversely affected the rights, safety, or welfare of the subjects or others, or substantially compromised the research data.

All adverse events that do not meet any of the criteria for serious, should be regarded as **non-serious adverse events**.

#### 11.1.4 Adverse Event Reporting Period

For this study, the follow-up period is defined as up to 10 minutes after arrival to PACU or TOF ratio is > 0.9 (whichever occurs first).

#### 11.1.5 Preexisting Condition

A preexisting condition is one that is present at the start of the study. A preexisting condition should be recorded as an adverse event if the frequency, intensity, or the character of the condition worsens during the study period.

#### 11.1.6 Post-study Adverse Event

All unresolved adverse events should be followed by the sponsor-investigator until the events are resolved, the subject is lost to follow-up, or the adverse event is otherwise explained. At the last scheduled visit, the sponsor-investigator should instruct each subject to report, to the sponsor-investigator, any subsequent event(s) that the subject, or the subject's personal physician, believes might reasonably be related to participation in this study.

#### 11.1.7 Hospitalization, Prolonged Hospitalization or Surgery

Any adverse event that results in hospitalization or prolonged hospitalization should be documented and reported as a serious adverse event unless specifically instructed otherwise in this protocol. Any condition responsible for surgery should be documented as an adverse event if the condition meets the criteria for an adverse event.

Neither the condition, hospitalization, prolonged hospitalization, nor surgery are reported as an adverse event in the following circumstances:

 Hospitalization or prolonged hospitalization for therapy of the target disease of the study, unless it is a worsening or increase in frequency of hospital admissions as judged by the clinical investigator.

#### 11.2 Recording of Adverse Events

At each contact with the subject, the study team must seek information on adverse events by specific questioning and, as appropriate, by examination. Information on all adverse events should be recorded immediately in the source document, and also in the appropriate adverse event section of the electronic case report form (CRF). All clearly related signs, symptoms, and abnormal diagnostic, laboratory or procedure results should recorded in the source document.

All adverse events occurring during the study period must be recorded. The clinical course of each event should be followed until resolution, stabilization, or until it has been ultimately determined that the study treatment or participation is not the probable cause. Serious adverse events that are still ongoing at the end of the study period must be followed up, to determine the final outcome. Any serious adverse event that occurs during the Adverse Event Reporting Period and is considered to be at least possibly related to the study treatment or study participation should be recorded and reported immediately.

## 11.3 Reporting of Serious Adverse Events and Unanticipated Problems

When an adverse event has been identified, the study team will take appropriated action necessary to protect the study participant and then complete the Study Adverse Event Worksheet and log. The sponsor-investigator will evaluate the event and determine the necessary follow-up and reporting required.

## 11.3.1 Sponsor-Investigator reporting: notifying the Mayo IRB

The sponsor-investigator will report to the Mayo IRB any UPIRTSOs and Non-UPIRTSOs according to the Mayo IRB Policy and Procedures. Each participating site will report SAEs to their respective IRB or Ethics Committee with copy of submission and review provided to the leading site. Should there be any SAEs at any of the participating sites; the study team at that site will notify the primary site (Mayo Clinic in Florida) within 24 hours of learning of the event.

Any serious adverse event (SAE) which the Principal Investigator has determined to be a UPIRTSO will be reported to the Mayo IRB as soon as possible but no later than 5 working days after the investigator first learns of the problem/event.

The following information will be collected on the adverse event worksheet (and entered in the research database):

- Study ID
- Disease
- The date the adverse event occurred
- Description of the adverse event
- Relationship of the adverse event to the research device\*
- Determination if the adverse event was expected
- The severity of the adverse event (severity scale described below \*\*)
- If any intervention was necessary
- Resolution (was the incident resolved spontaneously, or after discontinuing treatment)

#### • Date of Resolution

The sponsor-investigator will review all adverse event reports to determine if specific reports need to be made to the IRB. The sponsor-investigator will sign and date the adverse event report when it is reviewed. For this protocol, only directly related SAEs/UPIRTSOs will be reported to the IRB.

# \* Relationship Index

The relationship of an AE to the Investigational Device is a clinical decision by the sponsor-investigator (PI) based on all available information at the time of the completion of the eCRF and is graded as follows:

- 1. Not related: a reaction for which sufficient information exists to indicate that the etiology is unrelated to the use and proper application of study device.
- 2. Unlikely: a clinical event, including laboratory test abnormality, with a temporal relationship to use of the study device which makes a causal relationship improbable and in which use of other devices, chemicals, or underlying disease provide plausible explanations.
- 3. Possible: a clinical event, including laboratory test abnormality, with a reasonable time sequence to use of the study device but which could also be explained by concurrent disease or use of other devices or chemicals.
- 4. Probable: a clinical event including laboratory test abnormality, with a reasonable time sequence to use of the study device, unlikely to be attributed to concurrent disease or use of other devices or chemicals.
- 5. Definite: a reaction that follows a reasonable temporal sequence from the use of the study device.

## \*\* Severity Scale

The maximum intensity of an AE during a day should be graded according to the definitions below and recorded in details as indicated on the CRF. If the intensity of an AE changes over a number of days, then separate entries should be made having distinct onset dates.

- 1. Mild: AEs are usually transient, requiring no special treatment, and do not interfere with patient's daily activities.
- 2. Moderate: AEs typically introduce a low level of inconvenience or concern to the patient and may interfere with daily activities, but are usually ameliorated by simple therapeutic measures.

3. Severe: AEs interrupt a patient's usual daily activity and traditionally require systemic drug therapy or other treatment.

## 11.4 Medical Monitoring

It is the responsibility of the Principal Investigator to oversee the safety of the study at his/her site. This safety monitoring will include careful assessment and appropriate reporting of adverse events as noted above, as well as the construction and implementation of a site data and safety-monitoring plan (see section 10 "Study Monitoring, Auditing, and Inspecting"). Medical monitoring will include a regular assessment of the number and type of serious adverse events.

# 12 Data Handling and Record Keeping

## **12.1** Confidentiality

Information about study subjects will be kept confidential and managed according to the requirements of the Health Insurance Portability and Accountability Act of 1996 (HIPAA). Those regulations require a signed subject authorization informing the subject of the following:

- What protected health information (PHI) will be collected from subjects in this study
- Who will have access to that information and why
- Who will use or disclose that information
- The rights of a research subject to revoke their authorization for use of their PHI.

In the event that a subject revokes authorization to collect or use PHI, the investigator, by regulation, retains the ability to use all information collected prior to the revocation of subject authorization. For subjects that have revoked authorization to collect or use PHI, attempts should be made to obtain permission to collect at least vital status (long term survival status that the subject is alive) at the end of their scheduled study period.

#### 12.2 Source Documents

Source data is all information, original records of clinical findings, observations, or other activities in a clinical trial necessary for the reconstruction and evaluation of the trial. Source data are contained in source documents. Examples of these original documents and data records include: hospital records and any forms completed specifically for this study.

#### 12.3 Case Report Forms

All data necessary for this study will be obtained from EHR or at the time devices are being used and recorded on the electronic Case Report Forms (CRFs) created in REDCap. All missing data will be explained.

#### 12.4 Data Management

Study data to be collected and managed using EHR and study-generated source documents and transcribed into electronic CRFs in REDCap, electronic data capture software, hosted by CTSA

at Mayo Clinic. REDCap (Research Electronic Data Capture) is a secure, web-based application designed to support data capture for research studies, providing 1) an intuitive interface for validated data entry; 2) audit trails for tracking data manipulation and export procedures; 3) automated export procedures for seamless data downloads to common statistical packages; and 4) procedures for importing data from external sources.

#### 12.5 Data Processing

All study date will be stored and analyzed at Mayo Clinic in Florida using the REDCap electronic data capture tool.

#### 12.6 Data Security and Confidentiality

All source documents including clinical findings, observations or other activities will be stored in a REDCap database that will be designed by an Investigator. Access to the REDCap database will be limited to the Principal Investigator, Investigators, Study Team members, and Statistician.

#### 12.7 Data Quality Assurance

Once the study is completed the Principal Investigator will randomly select 3 participants and compare the data documented in the EHR with what is entered into the REDCap database. If there is any discrepancy, the Principal Investigator and/or Investigators will cross-reference all 100 patients to ensure accuracy.

#### 12.8 Data Clarification Process

For any data query the Principal Investigator and Investigators will meet to clarify the data queried and make corrections based on consensus.

#### 12.9 Records Retention

The sponsor-investigator will maintain records and essential documents related to the conduct of the study. These will include subject case histories and regulatory documents. Principal Investigator will maintain regulatory and essential study documents to ensure compliance with local and federal policies/guidelines.

The sponsor-investigator will retain the specified records and reports:

 As outlined in the Mayo Clinic Research Policy Manual –"Retention of and Access to Research Data Policy"

# 13 Study Monitoring, Auditing, and Inspecting

#### 13.1 Study Monitoring Plan

The investigator will allocate adequate time for such monitoring activities. The Investigator will also ensure that the compliance or quality assurance reviewer is given access to all the study-related documents.

#### 13.2 Auditing and Inspecting

The investigator will permit study-related monitoring, audits, and inspections by the IRB, the sponsor, and government regulatory agencies, of all study related documents (e.g. source documents, regulatory documents, data collection instruments, study data etc.).

Participation as an investigator in this study implies acceptance of potential inspection by government regulatory authorities and applicable compliance offices.

#### 14 Ethical Considerations

This study is to be conducted according to United States and International government regulations and Institutional research policies and procedures.

This protocol and any amendments will be submitted to a properly constituted local Institutional Review Board (IRB), in agreement with local legal prescriptions, for formal approval of the study. The decision of the IRB concerning the conduct of the study will be made in writing to the sponsor-investigator before commencement of this study.

All subjects for this study will be provided a consent form describing this study and providing sufficient information for subjects to make an informed decision about their participation in this study. This consent form will be submitted with the protocol for review and approval by the IRB for the study. The formal consent of a subject, using the Approved IRB consent form, must be obtained before that subject undergoes any study procedure. The consent form must be signed by the subject and the individual obtaining the informed consent.

# 15 Study Finances

#### 15.1 Funding Source

This investigator initiated study is not funded. Study coordinator's time is supported by the Department of Anesthesiology and funding for statistical analysis will be provided from the Principal Investigator's research fund.

#### 15.2 Conflict of Interest

Any study team member who has a conflict of interest with this study (patent ownership, royalties, or financial gain greater than the minimum allowable by their institution, etc.) must have the conflict reviewed by a properly constituted Conflict of Interest Committee with a Committee-sanctioned conflict management plan that has been reviewed and approved by the study sponsor-investigator prior to participation in this study.

No financial conflicts of interested are anticipated or have been identified for this study.

# 15.3 Subject Stipends or Payments

No payment is given to study participants.

#### 16 Publication Plan

The primary responsibility for publication of the study results is with the Primary Investigator. After the complication of study and prior to publication, the study results will be shared with all Investigators. The study will be registered at ClinicalTrials.gov prior to subject recruitment along with the posting of the results within 12 months of final data collection for the primary outcome measure.

#### 17 References

- Berg, H., J. Roed, J. Viby-Mogensen, C. R. Mortensen, J. Engbaek, L. T. Skovgaard, and J. J. Krintel. 1997. 'Residual neuromuscular block is a risk factor for postoperative pulmonary complications. A prospective, randomised, and blinded study of postoperative pulmonary complications after atracurium, vecuronium and pancuronium', *Acta Anaesthesiol Scand*, 41: 1095-103.
- Cammu, G., J. De Witte, J. De Veylder, G. Byttebier, D. Vandeput, L. Foubert, G. Vandenbroucke, and T. Deloof. 2006. 'Postoperative residual paralysis in outpatients versus inpatients', *Anesth Analg*, 102: 426-9.
- Elyassi, A. R., and H. H. Rowshan. 2009. 'Perioperative management of the glucose-6-phosphate dehydrogenase deficient patient: a review of literature', *Anesth Prog*, 56: 86-91.
- Eriksson, L. I., E. Sundman, R. Olsson, L. Nilsson, H. Witt, O. Ekberg, and R. Kuylenstierna. 1997. 'Functional assessment of the pharynx at rest and during swallowing in partially paralyzed humans: simultaneous videomanometry and mechanomyography of awake human volunteers', *Anesthesiology*, 87: 1035-43.
- Evora, P. R., L. Alves Junior, C. A. Ferreira, A. C. Menardi, S. Bassetto, A. J. Rodrigues, A. Scorzoni Filho, and W. V. Vicente. 2015. 'Twenty years of vasoplegic syndrome treatment in heart surgery. Methylene blue revised', *Rev Bras Cir Cardiovasc*, 30: 84-92.
- Faber, P., A. Ronald, and B. W. Millar. 2005. 'Methylthioninium chloride: pharmacology and clinical applications with special emphasis on nitric oxide mediated vasodilatory shock during cardiopulmonary bypass', *Anaesthesia*, 60: 575-87.

Fortier, L. P., D. McKeen, K. Turner, E. de Medicis, B. Warriner, P. M. Jones, A. Chaput, J. F. Pouliot, and A. Galarneau. 2015. 'The RECITE Study: A Canadian Prospective, Multicenter Study of the Incidence and Severity of Residual Neuromuscular Blockade', *Anesth Analg*, 121: 366-72.

- Fuchs-Buder, T., C. Claudius, L. T. Skovgaard, L. I. Eriksson, R. K. Mirakhur, J. Viby-Mogensen, and Meeting th International Neuromuscular. 2007. 'Good clinical research practice in pharmacodynamic studies of neuromuscular blocking agents II: the Stockholm revision', *Acta Anaesthesiol Scand*, 51: 789-808.
- Grayling, M., and B. P. Sweeney. 2007. 'Recovery from neuromuscular blockade: a survey of practice', *Anaesthesia*, 62: 806-9.
- Kaisers, U., J. M. Langrehr, M. Haack, A. Mohnhaupt, P. Neuhaus, and R. Rossaint. 1995. 'Hepatic venous catheterization in patients undergoing positive end-expiratory pressure ventilation after OLT: technique and clinical impact', *Clin Transplant*, 9: 301-6.
- McCartney, S. L., L. Duce, and K. Ghadimi. 2018. 'Intraoperative vasoplegia: methylene blue to the rescue!', *Curr Opin Anaesthesiol*, 31: 43-49.
- Murphy, G. S., J. W. Szokol, M. J. Avram, S. B. Greenberg, J. H. Marymont, J. S. Vender, J. Gray, E. Landry, and D. K. Gupta. 2011. 'Intraoperative acceleromyography monitoring reduces symptoms of muscle weakness and improves quality of recovery in the early postoperative period', *Anesthesiology*, 115: 946-54.
- Murphy, G. S., J. W. Szokol, M. J. Avram, S. B. Greenberg, T. D. Shear, J. S. Vender, K. N. Parikh, S. S. Patel, and A. Patel. 2015. 'Residual Neuromuscular Block in the Elderly: Incidence and Clinical Implications', *Anesthesiology*, 123: 1322-36.
- Murphy, G. S., J. W. Szokol, J. H. Marymont, S. B. Greenberg, M. J. Avram, and J. S. Vender. 2008. 'Residual neuromuscular blockade and critical respiratory events in the postanesthesia care unit', *Anesth Analg*, 107: 130-7.
- Naguib, M., S. J. Brull, A. F. Kopman, J. M. Hunter, B. Fulesdi, H. R. Arkes, A. Elstein, M. M. Todd, and K. B. Johnson. 2018. 'Consensus Statement on Perioperative Use of Neuromuscular Monitoring', *Anesth Analg*, 127: 71-80.
- Naguib, M., A. F. Kopman, and J. E. Ensor. 2007. 'Neuromuscular monitoring and postoperative residual curarisation: a meta-analysis', *Br J Anaesth*, 98: 302-16.
- Naguib, M., A. F. Kopman, C. A. Lien, J. M. Hunter, A. Lopez, and S. J. Brull. 2010. 'A survey of current management of neuromuscular block in the United States and Europe', *Anesth Analg*, 111: 110-9
- Renew, J. R., and S. J. Brull. 2019. 'The RECITE-US study: Stacking the odds in a chronic patient safety threat', *J Clin Anesth*, 56: 132-33.
- Sundman, E., H. Witt, R. Olsson, O. Ekberg, R. Kuylenstierna, and L. I. Eriksson. 2000. 'The incidence and mechanisms of pharyngeal and upper esophageal dysfunction in partially paralyzed humans: pharyngeal videoradiography and simultaneous manometry after atracurium', *Anesthesiology*, 92: 977-84.
- Todd, M. M., and B. J. Hindman. 2015. 'The Implementation of Quantitative Electromyographic Neuromuscular Monitoring in an Academic Anesthesia Department: Follow-Up Observations', *Anesth Analg*, 121: 836-8.
- Todd, M. M., B. J. Hindman, and B. J. King. 2014. 'The implementation of quantitative electromyographic neuromuscular monitoring in an academic anesthesia department', *Anesth Analg*, 119: 323-31.
- Woehlck, H. J., B. T. Boettcher, K. K. Lauer, D. C. Cronin, J. C. Hong, M. A. Zimmerman, J. Kim, and M. Selim. 2016. 'Hydroxocobalamin for Vasoplegic Syndrome in Liver Transplantation: Restoration of Blood Pressure Without Vasospasm', *A A Case Rep*, 7: 247-50.

# 18 List of In-Text Tables

# 18.1 Schedule of Events

| | Schedule of Events | |
|-----------------------------|--------------------|---------|
| Study Activity | Visit 1 | Visit 2 |
| Tetragraph | | X |
| Informed consent | X | |
| Review of Medical<br>Record | X | |
| Adverse event evaluation | | Х |

# 18.2 Intraoperative Data

| Study ID: | | | | | |
|---|---|---|---|---|---|
| Examiner Initials: | | | Date (dd / mm / yyyy): | | |
| Muscle relaxant na | Muscle relaxant name: | | | | |
| Muscle relaxant total dose (mg): | | | | | |
| Time of last muscl | e relaxant ( | lose (mm : hl | n): | : am / p | m |
| Reversal agent name: | | | | | |
| Reversal agent dos | se (mg): | | | | |

| Time of reversal as | gent | administration (mm : hh): | : | am / pm |
|---|---|---|---|---|
| Time of extubation | n: | : | am / pm | |
| TOF ratio / TOF co | ount | at the time of reversal (if av | ailable): | |
| Monitor used during reversal: PNS / TetraGraph / IntelliVue NMT / ToFscan / None | | | | |
| Site of monitoring during reversal: | | Hand / Face / Leg | | |
| TOF ratio / TOF count at the time of extubation (if available): | | | | |
| Monitor used at extubation: PNS / IntelliVue NMT / ToFscan / None | | | | |
| Site of monitoring: | | Hand / Face / Leg | | |

# 18.3 Monitoring data

| Study ID | | | | | |
|---|---|---|---|---|---|
| Date of Surgery (dd / mm / yyyy): | | | | | |
| Initials: Dominar | | nt side: | L / | R | Age (yrs): |
| Wrist circumference (right): | 1 | Vrist c | ircumferen | ce (left): | |
| Ankle circumference (right): | , | Ankle o | ircumferen | ce (left): | |
| Weight (kg): Height ( | cm): | | | BMI: | |

# TetraGraph (TG) Arm tested: dominant / non-dominant

| | Thumb | Toe | TOFR #3 (if needed) |
|---|---|---|---|
| Calibrated baseline<br>TOFR and supramax<br>current | | | |
| Time to TOFC=0 | | | |
| pre-SGX | | | |
| +20 sec | | | |
| +40 sec | | | |
| +60 sec | | | |
| +120 sec | | | |
| +140 sec | | | |
| +180 sec | | | |
| +200 sec | | | |
| +220 sec | | | |
| +240 sec | | | |

| +260 sec |
|---|
| TOFC or TOFR +280 sec |
| TOFC or TOFR +300 sec |
| TOFC or TOFR at extubation |
| Time to recovery following SGX (TOFR ≥0.9) (two consecutive measurements) |

# 19 List of In-Text Figures

# 19.1 TetraGraph

